CLINICAL TRIAL: NCT04480463
Title: A Phase III Randomized, Double-Masked, Parallel Group, Multicenter Study to Compare the Efficacy, Safety, Tolerability, Pharmacokinetics, and Immunogenicity Between SCD411 and Eylea® in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: A Study to Comparing SCD411 and Eylea® in Subjects With Wet Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sam Chun Dang Pharm. Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCD411-CP101; 2019-004132-37 (EudraCT Number)
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Wet Age-related Macular Degeneration; Neovascular Age-related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; Neovascular; Exudative
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the unmasked investigator involved in performing the IVT injections will be unmasked to study treatment. These individuals are not allowed to discuss treatment and/or subject outcome with masked study staff, including the evaluating investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SCD411 (Experimental)
  Interventions: Drug: SCD411
- Aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: SCD411 — IVT (intravitreal) injection
  Arms: SCD411
Drug: Aflibercept — IVT injection
  Other Names: Eylea®
  Arms: Aflibercept

SUMMARY:
Age-related macular degeneration (AMD) is a leading cause of vision loss in adults. Abnormal blood vessels grow under the macula at the back of the eye, and also leak blood and fluid, which damages and scars the macula, affecting vision. The current standard of care for patients with neovascular (exudative / wet) AMD is anti-vascular endothelial growth factor (anti-VEGF) therapy, which prevents or slows down the growth of the abnormal blood vessels. SCD411 is being developed as a biosimilar to the reference product Eylea® (aflibercept), an anti-VEGF drug. The study aims to prove equivalence of SCD411 to Eylea in adults with wet AMD, and will look at safety, tolerance, effectiveness, immune response and the movement of the drug through the body.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent.
* Clinical diagnosis of wet (neovascular) age-related macular degeneration (AMD).
* BCVA (best corrected visual acuity) letter score of 73 to 35 at screening and prior to randomization. In addition, fellow eye should not be less than 35 letter score using the ETDRS chart or 2702 series number chart.
* Women of child-bearing potential with negative serum pregnancy test at screening must agree to use protocol-defined methods of contraception throughout study until 3 months after last injection of aflibercept/SCD411.
* Males with female partners of child-bearing potential must agree to use protocol-defined methods of contraception and refrain from donating sperm throughout study until 3 months after last injection of aflibercept/SCD411.

Exclusion Criteria:

* Any prior eye (study eye and fellow eye) or systemic treatment or surgery for neovascular AMD, except dietary supplements or vitamins.
* Any prior or current treatment with another investigational agent to great neovascular AMD in the study eye, except dietary supplements or vitamins.
* Fellow eye shows signed of AMD that may need treatment during study period.
* Any prior treatment with anti-VEGF agents in both eyes.
* Total lesion size >30.5 mm2, Blood, scars, atrophy, fibrosis, and neovascularization, based on assessment at screening.
* Central retina thickness of <300 µm in the study eye.
* Subretinal hemorrhage that is either 50% or more of the total lesion area.
* Scar or fibrosis making up >50% of the total lesion.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macular in the study eye.
* Cataract in the study eye that have Lens Opacity Classification System II (LOCS II) grade IV cataract in the study eye or in the Investigator's opinion, interferes with visualization of retina or retinal imaging.
* Inflammation outside the eyeball in either eye, or within the eyeball of the study eye.
* History of any vitreous hemorrhage in the study eye.
* History or clinical evidence of diabetic retinopathy, diabetic macular edema, or any other vascular disease.
* History of, treatment or surgery for detached retina.
* History of uncomplicated surgery within the eyeball or around the study eye, except lid surgery.
* Absence of lens in study eye.
* Uncontrolled hypertension, defined as systolic blood pressure (BP) >160 mmHg or diastolic BP >100 mmHg under appropriate antihypertensive treatment.
* Hypersensitivity to aflibercept or medications used in the study (fluorescein, mydriatic eye drops, etc.).
* Pregnancy or lactation at Screening or at baseline for women of child-bearing potential.
* History of blood clotting events.
* History or evidence of cardiac conditions, or inability to perform any physical activity without discomfort; ventricular arrhythmia; and atrial fibrillation.
* History of laser therapy in the macular region.
* Any prior or current treatment with corticosteroids inside or immediately around the study eye.
* Any prior or current treatment involving the macula with photodynamic therapy (PDT) with verteporfin, transpupillary thermotherapy, radiation therapy, or retinal laser treatment in the study eye.
* Any prior or current treatment with pan-retinal photocoagulation.
* Any prior or current treatment with ethambutol; deferoxamine and topiramate; tamoxifen, hydroxychloroquine, chloroquine, or vigabatrin; and amiodarone.
* Any investigational product for the treatment of eye conditions and systemic conditions, 30 days or 5 half-lives (whichever is longer), prior to randomization, and throughout the study, except dietary supplements or vitamins.
* Intraocular pressure ≥25 mmHg in spite of anti-glaucoma treatment.
* Any prior or ongoing systemic medical condition (including but not limited to infectious, inflammatory, psychiatric, neurological, renal, hepatic, respiratory conditions or malignancies) or clinically significant screening laboratory value that in the opinion of the investigator may present a safety risk, interfere with study compliance and follow-up, or confound data interpretation throughout the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byung Jhip Ha, Study Director — Sam Chun Dang Pharm. Co. Ltd.
Locations (99):
- United States (12):
  - SCD Research Site, Campbell, California
  - SCD Research Site, Clearwater, Florida
  - SCD Research Site, Coral Springs, Florida
  - SCD Research Site, Fort Myers, Florida
  - SCD Research Site, Stuart, Florida
  - SCD Research Site, Marietta, Georgia
  - SCD Research Site, Lemont, Illinois
  - SCD Research Site, Liverpool, New York
  - SCD Research Site, Springfield, Oregon
  - SCD Research Site, Rapid City, South Dakota
  - SCD Research Site, Abilene, Texas
  - SCD Research Site, Willow Park, Texas
- Australia (4):
  - SCD Research Site, Liverpool, New South Wales
  - SCD Research Site, Sydney, New South Wales
  - SCD Research Site, East Melbourne, Victoria
  - SCD Research Site, Nedlands, Western Australia
- Bulgaria (2):
  - SCD Research Site, Sofia, Sofia-Grad
  - SCD Research Site, Sofia
- Czechia (2):
  - SCD Research Site, Pardubice, Pardubický kraj
  - SCD Research Site, Prague
- Hungary (4):
  - SCD Research Site, Budapest
  - SCD Research Site, Debrecen
  - SCD Research Site, Nyíregyháza
  - SCD Research Site, Pécs
- India (6):
  - SCD Research Site, Wardha, Maharashtra
  - SCD Research Site, Bhubaneswar, Odisha
  - SCD Research Site, Jaipur, Rajasthan
  - SCD Research Site, Hyderabad, Telangana
  - SCD Research Site, Lucknow, Uttar Pradesh
  - SCD Research Site, Kolkata, West Bengal
- Israel (11):
  - SCD Research Site, Haifa
  - SCD Research Site, Holon
  - SCD Research Site, Jerusalem
  - SCD Research Site, Kfar Saba
  - SCD Research Site, Nahariya
  - SCD Research Site, Petah Tikva
  - SCD Research Site, Ramat Gan
  - SCD Research Site, Rehovot
  - SCD Research Site, Tel Aviv
  - SCD Research Site, Tiberias
  - SCD Research Site, Ẕerifin
- Japan (22):
  - SCD Research Site, Nagoya, Aiti
  - SCD Research Site, Kurume, Hukuoka
  - SCD Research Site, Amagasaki, Hyôgo
  - SCD Research Site, Kobe, Hyōgo
  - SCD Research Site, Nishinomiya, Hyōgo
  - SCD Research Site, Kagoshima, Kagoshima-ken
  - SCD Research Site, Kyoto, Kyôto
  - SCD Research Site, Nakagami, Okinawa
  - SCD Research Site, Chuo Ku, Tokyo
  - SCD Research Site, Hachiōji, Tokyo
  - SCD Research Site, Meguro City, Tokyo
  - SCD Research Site, Nerima-ku, Tokyo
  - SCD Research Site, Ube, Yamaguchi
  - SCD Research Site, Fukuoka
  - SCD Research Site, Fukushima
  - SCD Research Site, Kita-ku
  - SCD Research Site, Nagakute
  - SCD Research Site, Niigata
  - SCD Research Site, Saga
  - SCD Research Site, Sakai
  - SCD Research Site, Sakura
  - SCD Research Site, Toyama
- Latvia (2):
  - SCD Research Site, Jelgava
  - SCD Research Site, Riga
- Poland (10):
  - SCD Research Site, Wałbrzych, Lower Silesian Voivodeship
  - SCD Research Site, Wroclaw, Lower Silesian Voivodeship
  - SCD Research Site, Warsaw, Masovian Voivodeship
  - SCD Research Site, Rzeszów, Podkarpackie Voivodeship
  - SCD Research Site, Gdansk, Pomeranian Voivodeship
  - SCD Research Site, Katowice, Silesian Voivodeship
  - SCD Research Site, Olsztyn, Warminsko-marzurskie
  - SCD Research Site, Bydgoszcz
  - SCD Research Site, Lublin
  - SCD Research Site, Warsaw
- Russia (2):
  - SCD Research Site, Moscow
  - SCD Research Site, Novosibirsk
- Slovakia (4):
  - SCD Research Site, Bratislava
  - SCD Research Site, Poprad
  - SCD Research Site, Trebišov
  - SCD Research Site, Žilina
- South Korea (11):
  - SCD Research Site, Guri-si, Gyeonggido
  - SCD Research Site, Suwon, Gyeonggido
  - SCD Research Site, Changwon-Si, Gyeongsangnam-do
  - SCD Research Site, Cheongju-si, North Chungcheong
  - SCD Research Site, Busan
  - SCD Research Site, Daegu
  - SCD Research Site, Daejeon
  - SCD Research Site, Gwangju
  - SCD Research Site, Incheon
  - SCD Research Site, Jinju
  - SCD Research Site, Seoul
- Spain (7):
  - SCD Research Site, Sant Cugat del Vallès, Barcelona
  - SCD Research Site, Barcelona
  - SCD Research Site, Bilbao
  - SCD Research Site, Majadahonda
  - SCD Research Site, Valencia
  - SCD Research Site, Valladolid
  - SCD Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: FDA Recalls, Market Withdrawals, and Safety Alerts — http://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCD411 | Aflibercept
Started | 288 | 288
Completed | 259 | 256
Not Completed | 29 | 32
Not completed — Death | 0 | 1
Not completed — Adverse Event | 6 | 8
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 2 | 5
Not completed — Decision by the sponsor or administrative decision for a reason other than that of an AE | 2 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Subject missed any of first 2 doses (IVT I injection of IP at Day 1 or Week 4) after randomization | 0 | 1
Not completed — A decrease in BCVA of ≥30 letters compared with the last assessment of VA | 1 | 0
Not completed — Subretinal hemorrhage involving center of fovea or, size of hemorrhage was ≥50% of total lesion area | 1 | 0
Not completed — Other | 6 | 4

BASELINE CHARACTERISTICS:
Population: Included all randomized subjects who received at least 1 injection of the IP. Numbers were based on planned treatment group. Two subjects met the exclusion criteria but were randomized in error; however, they did not receive any IP injection. A third subject also did not receive any IP injection. These 3 subjects were excluded from all analyses sets.
Groups:
- Total: Total of all reporting groups
Arm/Group | SCD411 | Aflibercept | Total
Number analyzed (Participants) | 287 | 286 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (8) | 73.6 (8.55) | 73.5 (8.27)
Age, Customized [Count of Participants; unit: Participants]
  50 to less than 65 years | 33 | 40 | 73
  65 to less than 75 years | 131 | 119 | 250
  Greater than or equal to 75 years | 123 | 127 | 250
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 147 | 296
  Male | 138 | 139 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 278 | 276 | 554
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 97 | 90 | 187
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 188 | 194 | 382
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 7 | 6 | 13
  Bulgaria | 2 | 2 | 4
  Czechia | 3 | 3 | 6
  Hungary | 22 | 17 | 39
  India | 8 | 1 | 9
  Israel | 42 | 42 | 84
  Japan | 30 | 30 | 60
  Latvia | 10 | 13 | 23
  Poland | 37 | 50 | 87
  South Korea | 59 | 59 | 118
  Russia | 12 | 10 | 22
  Slovakia | 16 | 13 | 29
  Spain | 20 | 24 | 44
  United States | 19 | 16 | 35
Weight [Mean (Standard Deviation); unit: kilograms] — Population: A subject from the SCD411 group had missing vital sign data (including body weight and height)
  kilograms
    number analyzed (Participants) | 286 | 286 | 572
    (all) | 72.39 (15.244) | 72.26 (12.280) | 72.32 (14.757)
Height [Mean (Standard Deviation); unit: centimeters] — Population: A subject from the SCD411 group had missing vital sign data (including body weight and height)
  centimeters
    number analyzed (Participants) | 286 | 286 | 572
    (all) | 164.02 (9.117) | 164.64 (8.976) | 164.33 (9.045)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: A subject from the SCD411 group had missing vital sign data (including body weight and height)
  kg/m^2
    number analyzed (Participants) | 286 | 286 | 572
    (all) | 26.81 (4.682) | 26.53 (4.154) | 26.67 (4.424)
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: Letters correctly read] | 58.6 (10.75) | 59.9 (10.60) | 59.3 (10.69)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA (Best Corrected Visual Acuity)
Description: Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) letters score or 2702 charts
Time Frame: Baseline to Week 8
Population: The Full Analysis Set included all randomized subjects who received at least 1 injection of the study drug.
Measure: Mean (95% Confidence Interval); unit: Letters correctly read
Arm/Group | SCD411 | Aflibercept
Number analyzed (Participants) | 287 | 286
Letters correctly read | 5.5 [4.5 to 6.5] | 5.9 [4.8 to 6.9]

2. Secondary Outcome: Change From Baseline in BCVA (Best Corrected Visual Acuity)
Description: Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) letters score or 2702 charts
Time Frame: Baseline to Week 52
Population: The Full Analysis Set included all randomized subjects who received at least 1 injection of the study drug.
Measure: Mean (95% Confidence Interval); unit: Letters correctly read
Arm/Group | SCD411 | Aflibercept
Number analyzed (Participants) | 287 | 286
Letters correctly read | 9.0 [7.6 to 10.4] | 7.7 [6.3 to 9.1]

3. Secondary Outcome: Percentage of Subjects With Anti-SCD411 Antibodies
Description: Assessed by blood samples
Time Frame: Baseline, Weeks 4, 8, 20, 36 and 52
Population: The Safety Set included all subjects who received at least 1 injection of the study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | SCD411
Number analyzed (Participants) | 287
Percentage of participants
  Baseline : Positive: number analyzed (Participants) | 281
  Baseline : Positive | 7.1
  Baseline : Negative: number analyzed (Participants) | 281
  Baseline : Negative | 92.9
  Week 4 : Positive: number analyzed (Participants) | 272
  Week 4 : Positive | 29.4
  Week 4 : Negative: number analyzed (Participants) | 272
  Week 4 : Negative | 70.6
  Week 8 : Positive: number analyzed (Participants) | 270
  Week 8 : Positive | 40.0
  Week 8 : Negative: number analyzed (Participants) | 270
  Week 8 : Negative | 60.0
  Week 20 : Positive: number analyzed (Participants) | 260
  Week 20 : Positive | 39.6
  Week 20 : Negative: number analyzed (Participants) | 260
  Week 20 : Negative | 60.4
  Week 36 : Positive: number analyzed (Participants) | 253
  Week 36 : Positive | 22.9
  Week 36 : Negative: number analyzed (Participants) | 253
  Week 36 : Negative | 77.1
  Week 52 : Positive: number analyzed (Participants) | 252
  Week 52 : Positive | 20.2
  Week 52 : Negative: number analyzed (Participants) | 252
  Week 52 : Negative | 79.8

ADVERSE EVENTS:
Time Frame: Adverse events were assessed beginning at enrollment (date of signed informed consent) and up to 28 days after the last dose of the study drug, up to Day 365.
Arm/Group | SCD411 | Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/287 | 1/286
Serious Adverse Events (participants affected / at risk) | 32/287 | 30/286
Other Adverse Events (participants affected / at risk) | 128/287 | 121/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SCD411 (N=287) | Aflibercept (N=286)
Visual acuity reduced (Eye disorders) | 2 | 1 — Study Eye
Retinal pigment epithelial tear (Eye disorders) | 2 | 0 — Study Eye
Amaurosis fugax (Eye disorders) | 0 | 1 — Study Eye
Retinal haemorrhage (Eye disorders) | 0 | 1 — Study Eye
Endophthalmitis (Infections and infestations) | 1 | 0 — Study Eye
Visual acuity reduced (Eye disorders) | 0 | 1 — Fellow eye
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 0
Aspergilloma (Infections and infestations) | 0 | 1
Bone tuberculosis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Venom poisoning (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
High-grade B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SCD411 (N=287) | Aflibercept (N=286)
Angina pectoris (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 3
Age-related macular degeneration (Eye disorders) | 2 | 3 — Fellow Eye
Blepharitis (Eye disorders) | 1 | 3 — Study Eye
Blepharitis (Eye disorders) | 1 | 3 — Fellow Eye
Cataract (Eye disorders) | 5 | 4 — Study Eye
Cataract (Eye disorders) | 3 | 3 — Fellow Eye
Conjunctival haemorrhage (Eye disorders) | 8 | 6 — Study Eye
Conjunctival haemorrhage (Eye disorders) | 3 | 1 — Fellow Eye
Corneal erosion (Eye disorders) | 0 | 4 — Study Eye
Dry eye (Eye disorders) | 5 | 4 — Study Eye
Dry eye (Eye disorders) | 5 | 4 — Fellow Eye
Eye pain (Eye disorders) | 3 | 3 — Study Eye
Lacrimation increased (Eye disorders) | 3 | 1 — Study Eye
Neovascular age-related macular degeneration (Eye disorders) | 5 | 4 — Study Eye
Neovascular age-related macular degeneration (Eye disorders) | 20 | 13 — Fellow Eye
Ocular hypertension (Eye disorders) | 0 | 3 — Study Eye
Posterior capsule opacification (Eye disorders) | 4 | 1 — Study Eye
Punctate keratitis (Eye disorders) | 3 | 2 — Study Eye
Retinal haemorrhage (Eye disorders) | 1 | 4 — Study Eye
Subretinal fluid (Eye disorders) | 3 | 1 — Study Eye
Visual acuity reduced (Eye disorders) | 11 | 12 — Study Eye
Visual impairment (Eye disorders) | 4 | 1 — Study Eye
Visual impairment (Eye disorders) | 3 | 0 — Fellow Eye
Vitreous detachment (Eye disorders) | 0 | 4 — Study Eye
Vitreous floaters (Eye disorders) | 5 | 3 — Study Eye
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Gastritis (Gastrointestinal disorders) | 1 | 4
Inguinal hernia (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
COVID-19 (Infections and infestations) | 16 | 21
Conjunctivitis (Infections and infestations) | 3 | 3 — Study Eye
Conjunctivitis (Infections and infestations) | 7 | 2 — Fellow Eye
Gastroenteritis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1
Sinusitis (Infections and infestations) | 4 | 1
Tooth abscess (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 10 | 7
Intraocular pressure increased (Investigations) | 5 | 3 — Study Eye
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypertension (Vascular disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04480463/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT04480463/SAP_001.pdf